CLINICAL TRIAL: NCT01427829
Title: Computer-assisted Psychosocial Risk Assessment (CaPRA) for Refugee Health and Settlement - Evaluation Phase
Brief Title: Computer-assisted Psychosocial Risk Assessment (CaPRA) for Refugee Health and Settlement
Acronym: CaPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FA-25340
Record Dates: First submitted 2011-08-22; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Computer; Screening; Decision Support System; Primary Care; Psychosocial; Refugees
Keywords: pilot; randomized controlled trial; RCT; computer; screening; community heath center; psychosocial; immigrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (CaPRA) (Experimental)
  Interventions: Behavioral: Computer-assisted Psychosocial Risk Assessment (CaPRA)
- Control (usual care) (No Intervention)
  Interventions: Behavioral: Computer-assisted Psychosocial Risk Assessment (CaPRA)

INTERVENTIONS:
Behavioral: Computer-assisted Psychosocial Risk Assessment (CaPRA) — The study intervention was a touch-screen self-assessment survey which eligible patients completed on a touch-screen iPad in Dari/Farsi language while waiting to see their medical practitioner. The Computer-assisted Psychosocial Risk Assessment (CaPRA) survey had questions on psychosocial risks (e.g., alcohol, tobacco and street drug use, sexual health, personal violence, post-traumatic stress disorder, depression, and food insecurity), cardiovascular risks (e.g., physical activity, weight, diabetes, and hypertension), road and home safety, stress buffers (e.g., coping and social support) and sociodemographics. The tool generated two tailored print-outs at the point of care. The recommendation sheet for patients summarized their disclosed risks in simple Dari/Farsi language along with contacts of relevant services. The risk-report for medical practitioner summarized patients' risks with possible referrals. This was attached to the medical chart prior to the consult.

SUMMARY:
The purpose of this study was to examine preliminary effect of Computer-assisted Psychosocial Risk Assessment tool (CaPRA) among Afghan refugees visiting medical professionals (family physicians or nurse practitioners) at a Community Health Center. The investigators examined the tool's acceptability among patients and its impact on patient satisfaction and patient intention to visit a psychosocial counselor as a proxy of potential to integrate medical and social care.

DETAILED DESCRIPTION:
The recent waves of refugees to Canada belong to regions of prolonged conflict and, thus arrive in compromised state of mental, physical, and social health. This complexity asks for provision of integrated medical and social care to newly arrived refugees. With this aim, a university-community initiative developed a Computer-assisted Psychosocial Risk Assessment tool (CaPRA) in Dari/Farsi for Afghan refugees. This innovative eHealth approach is first of its kind for Canadian refugees accessing primary care. In this model of care, patients complete an interactive multi-risk iPad computer survey in their own language before seeing the provider. The computer then generates individualized recommendation sheet for patients and a risk-report for providers at the point of care. The tool was developed through a collaborative process by working with Access Alliance Multicultural Health and Community Services and advisory board with community representatives.

ELIGIBILITY:
Inclusion Criteria:

* Afghan refugee patients
* Over 18 years of age
* Speak and read Dari /Farsi or English language
* Eligible for federal or provincial health care program
* Visiting a participating medical practitioner

Exclusion Criteria:

* Patient visiting a provider who has not consented for the study
* Patient accompanied by a family member for interpretation
* New patients
* Patients unable to receive study details due to logistical issue (e.g, no private room)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Patient intention to visit a psychosocial counselor | July to October post-visit
  Patients completed a paper-pencil Exit Survey in the intervention (CaPRA) and control (usual care) groups

SECONDARY OUTCOMES:
Patient satisfaction | July to October post-visit
  Patients completed a paper-pencil Exit Survey in the intervention (CaPRA) and control (usual care) groups
Patient acceptability | July to October post-visit
  Patients completed a paper-pencil Exit Survey in the intervention group (CaPRA)

CONTACTS AND LOCATIONS:
Overall Officials: Farah Ahmad, MBBS, MPH, PhD, Principal Investigator — University of Toronto / York University